CLINICAL TRIAL: NCT00289718
Title: Long-Term Persistence Follow-up Study to Evaluate the Immune Persistence of GSK Biologicals' Combined Hepatitis A / Hepatitis B Vaccine in Healthy Adult Volunteers
Brief Title: Long-Term Immune Persistence of GSK Biologicals' Combined Hepatitis A & B Vaccine Injected According to a 0,1,6 Month Schedule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 100556 (Y11); 100557 (Y12) (Other: GSK); 100558 (Y13) (Other: GSK); 100559 (Y14) (Other: GSK); 100560 (Y15) (Other: GSK)
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Results first posted 2010-08-26 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2016-11

CONDITIONS: Hepatitis B; Hepatitis A
Keywords: Combined Hepatitis A and B vaccine; Hepatitis A; Hepatitis B
MeSH Terms: conditions — Hepatitis B; Hepatitis A

ARMS (1):
- Twinrix Group (Experimental): Subjects who received 2 doses of Twinrix™ (lot A, B or C) in the primary study.
  As lot to lot consistency was assessed during the primary study, the 3 groups (lot A, B or C) were pooled into the Twinrix Group for data analyses during the long term follow-up.
  Interventions: Biological: Twinrix™ adult

INTERVENTIONS:
Biological: Twinrix™ adult — Intramuscular administration

SUMMARY:
The aim of this study is to evaluate the long-term persistence of hepatitis A and B antibodies at Years 11, 12, 13, 14 and 15 years after subjects received their first dose of a 3 dose vaccination schedule of combined hepatitis A/hepatitis B vaccine. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

This protocol posting deals with objectives & outcome measures of the extension phase at year 11 to 15.

DETAILED DESCRIPTION:
This is a long-term follow-up study at Years 11, 12, 13, 14 and 15 after primary vaccination with GSK Biologicals' hepatitis A/hepatitis B vaccine (three-dose schedule, 3 different lots). To evaluate the long-term antibody persistence, volunteers will be bled at Years 11, 12, 13, 14 and 15 after the first vaccine dose of the primary vaccination course to determine their anti-HAV and anti-HBs antibody concentrations.

No additional subjects will be recruited during the course of this long-term study.

If a subject has become seronegative for anti-HAV antibodies or lost anti-HBs seroprotection concentrations at the long-term blood sampling time point (i.e. Years 11, 12, 13, 14 or 15), he/ she will be offered an additional vaccine dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects participating in this study should have received three-dose primary vaccination with combined hepatitis A/hepatitis B vaccine in the primary study.
* Written informed consent will be obtained from each subject before the blood sampling visit of each year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2004-11-01; Primary Completion 2005-03-02 (Actual); Study Completion 2005-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Van Damme P, Leroux-Roels G, Law B, Diaz-Mitoma F, Desombere I, Collard F, Tornieporth N, Van Herck K. Long-term persistence of antibodies induced by vaccination and safety follow-up, with the first combined vaccine against hepatitis A and B in children and adults. J Med Virol. 2001 Sep;65(1):6-13. PMID 11505437
- [Background] Van Damme P, Leroux-Roels G, Crasta P, Messier M, Jacquet JM, Van Herck K. Antibody persistence and immune memory in adults, 15 years after a three-dose schedule of a combined hepatitis A and B vaccine. J Med Virol. 2012 Jan;84(1):11-7. doi: 10.1002/jmv.22264. Epub 2011 Nov 3. PMID 22052690
- [Background] Van Herck K, Leroux-Roels G, Van Damme P, Srinivasa K, Hoet B. Ten-year antibody persistence induced by hepatitis A and B vaccine (Twinrix) in adults. Travel Med Infect Dis. 2007 May;5(3):171-5. doi: 10.1016/j.tmaid.2006.07.003. Epub 2006 Sep 20. PMID 17448944
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 100556 (Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100556 (Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 100556 (Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 100556 (Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 100556 are summarised with studies 100557, 100558, 100559, and 100560 on the GSK Clinical Study Register.
- Available data/document: Informed Consent Form: 100556 (Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Twinrix Group
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Twinrix Group
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (5.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Anti-hepatitis A Virus (Anti-HAV) Antibody Concentration
Description: Concentrations given as geometric mean concentration (GMC) expressed as milli-international unit per millilitre (mIU/mL).
Time Frame: At Years 11, 12, 13, 14, and 15 after the first vaccine dose of the 3-dose primary vaccination
Population: Analysis was performed on the Long Term According-to-Protocol (LT-ATP) cohort for immunogenicity, on subjects with available data for the defined timepoint
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Group
Number analyzed (Participants) | 33
mIU/mL
  Year 11 (N=33) | 369.1 [273.8 to 497.7]
  Year 12 (N=33) | 323.5 [233.8 to 447.7]
  Year 13 (N=32) | 293.7 [214.8 to 401.8]
  Year 14 (N=30) | 298.2 [217.0 to 409.6]
  Year 15 (N=29) | 274.4 [200.9 to 374.7]

2. Primary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed include pain, redness and swelling. Any was defined as occurrence of the specified solicited local symptom regardless of its intensity. Grade 3 pain was defined as pain that prevented normal everyday activities. Grade 3 swelling was greater than 100 millimeters (mm) i.e. >100mm.
Time Frame: During the 4-day (Day 0-3) follow-up period after additional HBV vaccination
Population: Analysis was performed on the Long Term Total cohort, on subjects who received an additional vaccine dose. Only 1 subject received an additional dose.
Measure: Number; unit: subjects
Groups:
- Twinrix Group: Subjects who received 2 doses of Twinrix™ (lot A) in the primary study.
Arm/Group | Twinrix Group
Number analyzed (Participants) | 1
subjects
  Pain | 1
  Redness | 0
  Swelling | 0

3. Primary Outcome: Number of Subjects Seropositive for Anti-HAV Antibodies
Description: A seropositive subject was defined as a vaccinated subject who had a anti-HAV antibody titres ≥ 33 mIU/ml.
Time Frame: At Years 11, 12, 13, 14, and 15 after the first vaccine dose of the 3-dose primary vaccination
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 33
Subjects
  Year 11 (N=33) | 33
  Year 12 (N=33) | 33
  Year 13 (N=32) | 32
  Year 14 (N=30) | 30
  Year 15 (N=29) | 29

4. Primary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentration
Description: Concentrations given as GMC expressed as mIU/mL. NOTE: There was a change of assay kit at Year 15 time-point, thus for the sake of bridging, blood samples corresponding to Year 14 were re-tested with ChemiLuminescence ImmunoAssay (CLIA). From Year 11 to Year 14, anti-HBs antibody concentrations were tested with ELISA with cut-off of 3.3 mIU/mL while, Year 14* onwards, anti-HBs antibody concentrations were tested with the CLIA with cut-off of 6.2 mIU/mL.
Time Frame: At Years 11, 12, 13, 14, and 15 after the first vaccine dose of the 3-dose primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Group
Number analyzed (Participants) | 33
mIU/mL
  Year 11 (N=33) | 123.6 [76.1 to 200.9]
  Year 12 (N=33) | 150.3 [92.9 to 243.0]
  Year 13 (N=32) | 77.8 [48.7 to 124.4]
  Year 14 (N=30) | 71.7 [45.5 to 113.1]
  Year 14* (N=28) | 95.3 [54.1 to 168.1]
  Year 15 (N=29) | 79.2 [45.7 to 137.3]

5. Primary Outcome: Number of Subjects Seropositive for Anti-HB Antibodies
Description: A seropositive subject was defined as a vaccinated subject who had anti-HB antibody titres ≥ 1 mIU/mL.
  NOTE: There was a change of assay kit at Year 15 time-point, thus for the sake of bridging, blood samples corresponding to Year 14 were re-tested with ChemiLuminescence ImmunoAssay (CLIA)
Time Frame: At Years 11, 12, 13, 14, and 15 after the first vaccine dose of the 3-dose primary vaccination
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | TWINRIX GROUP
Number analyzed (Participants) | 33
Subjects
  YEAR 11 (N=33) | 33
  YEAR 12 (N=33) | 33
  YEAR 13 (N=32) | 32
  YEAR 14 (N=30) | 29
  Year 14* (N=28) | 27
  YEAR 15 (N=29) | 28

6. Primary Outcome: Number of Subjects Seroprotected for Anti-HBs Antibodies.
Description: A seroprotected subject was defined as a subjects with the anti-HBs titres ≥ 10 mIU/mL.
  NOTE: There was a change of assay kit at Year 15 time-point, thus for the sake of bridging, blood samples corresponding to Year 14 were re-tested with ChemiLuminescence ImmunoAssay (CLIA)
Time Frame: At Years 11, 12, 13, 14, and 15 after the first vaccine dose of the 3-dose primary vaccination
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | TWINRIX GROUP
Number analyzed (Participants) | 33
Subjects
  YEAR 11 (N=33) | 33
  YEAR 12 (N=33) | 32
  YEAR 13 (N=32) | 32
  YEAR 14 (N=30) | 29
  Year 14* (N=28) | 27
  YEAR 15 (N=29) | 28

7. Primary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: A SAE was defined as any untoward medical occurrence that: resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the follow-up period after additional vaccination (minimum 30 days)
Population: as for outcome 2
Measure: Number; unit: subjects
Groups:
- Twinrix Group (Lot A): Subjects who received 2 doses of Twinrix™ (lot A) in the primary study.
- Twinrix Group (Lot B): Subjects who received 2 doses of Twinrix™ (lot B) in the primary study.
Arm/Group | Twinrix Group (Lot A) | Twinrix Group (Lot B)
Number analyzed (Participants) | 1 | 1
subjects | 0 | 1

8. Primary Outcome: Anti-Hepatitis B Surface Antigen (Anti-HBs) Antibody Concentration
Description: Concentrations given as GMC expressed as mIU/mL. If a subject became seronegative (< 10 mIU/mL) at any of the long-term blood sampling timepoint, he/she was offered an additional vaccine dose.
Time Frame: Before the additional dose and 1 month after the additional dose
Population: as for outcome 2
Measure: Number; unit: mIU/mL
Arm/Group | Twinrix Group
Number analyzed (Participants) | 1
mIU/mL
  before additional dose at Year 12 | 9.7
  1 month after additional dose at Year 12 | NA — One subject identified as eligible to receive the additional dose at Year 12 was withdrawn from the LT Cohort for immunogenicity because of non-compliance with the protocol therefore, blood sample was not taken
  before additional dose at Year 13 | 9.5
  1 month after additional dose at Year 13 | 15022.3

9. Primary Outcome: Number of Subjects Reporting Any Solicited General Symptoms.
Description: Solicited general symptoms assessed included fatigue, headache, malaise, nausea, vomiting and fever. Any was defined as any solicited general symptom reported irrespective of intensity and relationship to vaccination.
Time Frame: During the 4-day (Day 0-3) follow-up period after additional HBV vaccination
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 1
Subjects
  Any Fatigue | 0
  Any Headache | 0
  Any Malaise | 0
  Any Nausea | 0
  Any Vomiting | 0
  Any Fever | 0

10. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 30-day follow-up period after additional vaccination
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 1
subjects | 1

11. Primary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: as for outcome 7
Time Frame: At Years 11, 12, 13, 14, and 15 after the first vaccine dose of the 3-dose primary vaccination
Population: Analysis was performed on the LT Total Cohort that included all subjects who returned at a specified follow-up study and who belonged to the Total Cohort of the primary vaccination course.
Measure: Number; unit: Subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 51
Subjects | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs):Up to Year 15 and after additional HBV vaccination;Solicited local and general symptoms:During the 4-day follow-up period post additional dose;Unsolicited AEs:During the 30-day follow-up period post additional dose.
Description: Safety results were reported for subjects who received an additional vaccine dose. Only one subject received an additional dose
Arm/Group | Twinrix Group
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Twinrix Group (N=1)
Hallux valgus (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Twinrix Group (N=1)
Pain (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). The table shows updated results following complete retesting and reanalysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.